CLINICAL TRIAL: NCT01641991
Title: A Randomized Trial for the Assessment of Immunogenicity and Safety of Four Different Dosing Regimens of BioThrax® for Post-Exposure Prophylaxis for Anthrax in Adults
Brief Title: Assessment of the Immunogenicity and Safety of a Dose-Sparing BioThrax® AVA Schedule
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 11-0024; N01AI80006C
Record Dates: First submitted 2012-07-05; First posted 2012-07-17 (Estimated); Results first posted 2014-05-28 (Estimated); Last update posted 2014-05-28 (Estimated); Status verified 2014-04

CONDITIONS: Bacillus Anthracis (Anthrax)
Keywords: Bacillus anthracis, anthrax, vaccine, BioThrax®, dose-sparing
MeSH Terms: conditions — Anthrax | interventions — Biothrax

ARMS (4):
- Arm B: 0.50mL BioThrax® (Experimental): BioThrax® 0.50mL subcutaneously on Days 0, 28 and 0.50mL BioThrax® intramuscular 6 month boost; 75 subjects
  Interventions: Biological: BioThrax®
- Arm C: 0.50mL BioThrax® (Experimental): BioThrax® 0.50mL subcutaneously on Days 0, 14, 28 and 0.50mL BioThrax® intramuscular 6 month boost; 75 subjects
  Interventions: Biological: BioThrax®
- Arm D: 0.25mL BioThrax® (Experimental): BioThrax® 0.25mL subcutaneously on Days 0,14, and 28,and 0.50mL BioThrax® intramuscular 6 month boost; 75 subjects
  Interventions: Biological: BioThrax®
- Arm A: 0.50mL BioThrax® (Experimental): BioThrax® 0.50 ml subcutaneously on Days 0, 14, and 0.50mL BioThrax® intramuscular 6 month boost; 75 subjects
  Interventions: Biological: BioThrax®

INTERVENTIONS:
Biological: BioThrax® — BioThrax® is a sterile, milky white suspension made from cell free filtrates of microaerophilic cultures of an avirulent, nonencapsulated strain of Bacillus anthracis, will be administered as a 0.50mL IM injection 6 month boost for all groups
Biological: BioThrax® — BioThrax® will be administered as: Arm A: 0.50mL SC injection on Days 0 and 14; Arm B: 0.50mL SC injection on Days 0 and 28; Arm C: 0.50mL SC injection on Days 0, 14 and 28; Arm D: 0.25 mL SC injection on Days 0, 14 and 28.

SUMMARY:
A Phase IV, randomized, multicenter trial to assess the immunogenicity and safety of BioThrax® in varying dose regimens with the primary objective of obtaining information on possible dose-sparing strategies in the event of a major biothreat.

DETAILED DESCRIPTION:
This is a Phase IV, randomized, open-label immunogenicity and safety study to evaluate four dosing regimens of BioThrax® for Post-Exposure Prophylaxis (PEP) for anthrax. BioThrax® will be administered as a subcutaneous (SC) injection for the primary series and will be administered as an intramuscular (IM) injection for the boost. The four dosing regimens are: 0.50mL BioThrax® on Days 0, 14, and 6 month boost; 0.50mL BioThrax® on Days 0, 28 and 6 month boost; 0.50mL BioThrax® on Days 0, 14, 28 and 6 month boost and 0.25mL BioThrax® on Days 0, 14, and 28, 6 month boost with 0.50ml IM Approximately 300 subjects will be randomized 1:1:1:1 to one of the four study arms. Enrollment will be stratified by gender, with approximately equal numbers of males and females (18 through 65 years) enrolled into each dosing regimen. The Primary objective is to evaluate the immunogenicity of the four dosing regimens of BioThrax® using the Toxin Neutralization Assay (TNA). The secondary objective is to evaluate the safety of the four dosing regimens of BioThrax®.

ELIGIBILITY:
Inclusion Criteria:

* Subject able to provide informed consent;
* Female or male, 18 through 65 years of age, inclusive;
* If the subject is female and of childbearing potential, she agrees to practice abstinence from sexual intercourse with men (vaginal penetration by a penis, coitus) or use acceptable contraception, initiated at least 30 days prior to the first study vaccination through 56 days after the 6 month boost vaccination in order to avoid pregnancy:

  1. A woman is considered of childbearing potential unless post-menopausal (>/= 1 year without menses) or surgically sterilized (tubal ligation, bilateral oophorectomy, or hysterectomy)
  2. Acceptable contraception methods are restricted to effective devices (IUDs, NuvaRing®) or licensed hormonal products with use of method for a minimum of 30 days prior to vaccination, condoms with spermicidal agents, monogamous relationship with a vasectomized partner who has been vasectomized for 6 months or more prior to study entry, or successful Essure placement with documented confirmation test at least 3 months after the procedure, and any other Food and Drug Administration (FDA)-approved contraceptive method
* Be willing and able to return for all visits and blood collections for the duration of the study;
* Be able to understand and comply with planned study procedures;
* Agree to complete the memory aid and to report concomitant medications and Adverse Events during the study period.

Further clarification of inclusion/exclusion criteria:

Provided a subject meets all study inclusion criteria and none of the study exclusion criteria, the following conditions will not exclude the subject from study participation:

* History of gestational diabetes;
* Type II diabetes controlled with diet or oral hypoglycemic medications;
* Treated, controlled, uncomplicated hypertension;
* History of coronary artery disease, asymptomatic (New York Heart Association [NYHA] Function Class I), on a stable medical regimen. Persons meeting these criteria must be at least two years post-myocardial infarction, cardiac bypass surgery and/or percutaneous coronary interventions (e.g., angioplasty, stent placement) in order to qualify. Persons with a history of cardiac disease must be under the care of a physician;
* Cured, non-metastatic cancer (excluding hematologic malignancies), disease-free for five years;
* Localized skin cancer, resected (including squamous cell and basal cell carcinomas). Participants with a history of melanoma must be disease-free for five years;
* Exercise-induced bronchospasm controlled with inhaled medication(s) only;
* Mild asthma: Subjects who have not been hospitalized for asthma in the past two years and use only inhalers to control their symptoms will be eligible. Only low to medium doses of inhaled steroids, defined as </=3 puffs a day, are allowed. Persons who require oral or parenteral steroids will not be eligible.
* Subjects with isolated entrapment neuropathies, such as carpal tunnel syndrome, or compression neuropathies, such as lumbar radiculopathy, that are not associated with systemic disease or immune dysfunction may be eligible for enrollment. If the subject's condition has been stable for six months, surgery is not planned for the condition, the neurologic examination is normal (specifically no weakness or paresthesias), and the mononeuropathy will not interfere with the assessment of reactogenicity, the subject is eligible.
* Subjects with vitiligo who are otherwise healthy and the vitiligo is not widespread in the area of the vaccinations may be eligible for enrollment.
* Subjects with seasonal allergies are eligible provided the dose of nasal steroids that are used is < 800µg/day.

Exclusion Criteria:

* Have a prior history of anthrax or immunization against anthrax;
* Intend to enlist in the military during the study;
* Have a known allergy to aluminum hydroxide, formaldehyde, benzethonium chloride, or latex;
* (Females only) Be pregnant, plan to become pregnant at any time between the Screening Visit through 56 days after the 6 month boost vaccination, or refuse to use/not have used an acceptable method of birth control (see Inclusion Criterion 3) from 30 days prior to the first study vaccine dose through 56 days after the 6 month boost vaccination;
* Have received experimental products within 30 days before study entry or plan to receive experimental products at any time during the study;
* Have received a live vaccine within 30 days before study entry or plan to receive a live vaccine prior to Day 63 of the study or within 30 days of the 6 month boost;
* Have received an inactivated vaccine within 14 days before study entry or plan to receive an inactivated vaccine from Day 0 to Day 42 or within 14 days of the 6 month boost;
* Have received immunosuppressive therapy (including systemic steroids) within 3 months prior to study entry or plan to receive immunosuppressive therapy at any time during the study;
* Have received cytotoxic therapy in the previous 5 years or plan to receive cytotoxic therapy at any time during the study;
* Have received parenteral immunoglobulin or blood products within 3 months of the study or plan to receive parenteral immunoglobulin or blood products at any time during the study;
* Have a history of Guillain-Barré Syndrome;
* Have an active malignancy or history of metastatic or hematologic malignancy;
* Have Type I diabetes or Type II diabetes treated with insulin;
* Have cardiovascular disease (including any person with a history of cardiomyopathy or congestive heart failure);
* Have moderate to severe asthma, chronic obstructive pulmonary disease or other significant pulmonary disease;
* Have hepatic or renal insufficiency;
* Have an autoimmune, inflammatory, vasculitic or rheumatic disease including but not limited to systemic lupus erythematosus, polymyalgia rheumatica, rheumatoid arthritis or scleroderma;
* Have HIV, hepatitis B or hepatitis C infection;
* Have any other condition known to produce or be associated with immunosuppression;
* Have neuropathy or any other evolving neurological condition;
* Have an ongoing drug abuse/dependence (including alcohol) issues or a history of these issues within five years of enrollment;
* Have a seizure disorder;
* Have moderate or severe illness and/or an oral temperature >100.4 F within 3 days prior to vaccination;
* Have a blood pressure, heart rate or respiratory rate of Grade 2 or higher;
* Have any chronic condition that, in the opinion of the Investigator, would render vaccination unsafe or would interfere with study evaluations or completion of the study;
* Have a total White Blood Cell (WBC) count, Absolute Neutrophil Count (ANC), hemoglobin or platelet count that is Grade 2 or higher;
* Have a creatinine higher than the normal range;
* Have an Alanine Aminotransferase (ALT) of >/= 1.2 x Upper Limit of Normal;
* Have a value higher than trace for glucose and/or protein on urinalysis;
* Have a history of hospitalization for psychiatric illness, suicide attempt, or confinement for danger to self or others, within the past 10 years. (Subjects with a psychiatric disorder [not meeting exclusion criteria, e.g. attention-deficit hyperactivity disorder] that is controlled for a minimum of 3 months and the investigator has determined that the subject's mental status will not compromise the subject's ability to comply with protocol requirements may be enrolled);
* Be taking any of the following psychiatric drugs: aripiprazole, clozapine, ziprasidone, haloperidol, molindone, loxapine, thioridazine, thiothixene, pimozide, fluphenazine, risperidone, mesoridazine, quetiapine, trifluoperazine, trifluopromazine, chlorprothixene, chlorpromazine, perphenazine, olanzapine, carbamazepine, divalproex sodium, lithium carbonate or lithium citrate;
* Be taking more than one antidepressant drug not included in the list above (subjects taking only one antidepressant drug [not listed in excluded psychiatric drugs] who are stable for at least 3 months prior to enrollment without decompensating are allowed enrollment into the study provided the investigator determines the subject's mental status will not compromise the subject's ability to comply with protocol requirements);
* Have donated blood within 30 days of enrollment or plans to donate blood during the study.
* Have a tattoo in the area of the vaccination sites which will interfere with the assessment of injection site reactogenicity.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 328 (Actual)
Dates: Start 2012-07; Primary Completion 2013-03 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Emory Children's Center - Pediatric Infectious Diseases, Atlanta, Georgia
  - Cincinnati Children's Hospital Medical Center - Infectious Diseases, Cincinnati, Ohio
  - Baylor College of Medicine - Molecular Virology and Microbiology, Houston, Texas
  - Group Health Research Institute - Seattle, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were healthy adult males and females recruited from existing volunteer populations and from the communities at large around the clinical sites. Participants were enrolled and vaccinated between 05JUL2012 and 30NOV2012.
Groups:
- Arm A: 0.50mL BioThrax, Days 0, 14: BioThrax 0.50ml subcutaneously on Days 0, 14, and 0.50mL BioThrax intramuscularly at 6 month boost
- Arm B: 0.50mL BioThrax, Days 0, 28: BioThrax 0.50ml subcutaneously on Days 0, 28, and 0.50mL BioThrax intramuscularly at 6 month boost
- Arm C: 0.50mL BioThrax, Days 0, 14, 28: BioThrax 0.50ml subcutaneously on Days 0, 14, 28, and 0.50mL BioThrax intramuscularly at 6 month boost
- Arm D: 0.25mL BioThrax, Days 0, 14, 28: BioThrax 0.25ml subcutaneously on Days 0, 14, 28, and 0.50mL BioThrax intramuscularly at 6 month boost
Period: Overall Study
Arm/Group | Arm A: 0.50mL BioThrax, Days 0, 14 | Arm B: 0.50mL BioThrax, Days 0, 28 | Arm C: 0.50mL BioThrax, Days 0, 14, 28 | Arm D: 0.25mL BioThrax, Days 0, 14, 28
Started | 82 | 82 | 82 | 82
Completed | 73 | 74 | 65 | 66
Not Completed | 9 | 8 | 17 | 16
Not completed — Physician Decision | 0 | 1 | 7 | 5
Not completed — Withdrawal by Subject | 4 | 2 | 1 | 5
Not completed — Adverse Event | 2 | 1 | 2 | 1
Not completed — Lost to Follow-up | 0 | 2 | 3 | 1
Not completed — Protocol Violation | 1 | 1 | 3 | 0
Not completed — Pregnancy | 0 | 0 | 1 | 0
Not completed — no longer eligible | 2 | 1 | 0 | 4

BASELINE CHARACTERISTICS:
Population: All participants are included in the baseline analysis population.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A: 0.50mL BioThrax, Days 0, 14 | Arm B: 0.50mL BioThrax, Days 0, 28 | Arm C: 0.50mL BioThrax, Days 0, 14, 28 | Arm D: 0.25mL BioThrax, Days 0, 14, 28 | Total
Number analyzed (Participants) | 82 | 82 | 82 | 82 | 328
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.0 (10.8) | 36.7 (11.7) | 34.6 (11.5) | 36.5 (11.1) | 35.7 (11.2)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 82 | 82 | 82 | 82 | 328
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 42 | 40 | 41 | 166
  Male | 39 | 40 | 42 | 41 | 162
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 2 | 3 | 1 | 3 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 7 | 14 | 19 | 15 | 55
  White | 67 | 61 | 56 | 61 | 245
  More than one race | 6 | 3 | 5 | 2 | 16
  Unknown or Not Reported | 0 | 1 | 1 | 1 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 4 | 3 | 6 | 19
  Not Hispanic or Latino | 76 | 78 | 79 | 76 | 309
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 82 | 82 | 82 | 82 | 328

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Four-fold or Greater Increase From Baseline in Toxin Neutralization Antibody Assay (TNA) 50 Percent Neutralization Factor ( NF50 ) Antibody Titer
Description: Blood was collected from all participants prior to vaccination and at scheduled follow up visits weekly through Day 70, at Day 84 and at Day 100 for testing in the toxin neutralization antibody assay to determine the NF50 antibody titer. A participant met the threshold of a 4-fold rise in NF50 antibody titer if the post vaccination titer was an increase by 4-fold or more from the baseline (Day 0) titer.
Time Frame: Days 0, 7, 14, 21, 28 35, 42, 49, 56, 63, 70, 84 and 100
Population: The per protocol analysis population includes participants who met all inclusion and exclusion criteria, received all doses in the primary series, completed all scheduled visits up to and including the Day 100 visit in-window, and who contributed both pre- and post-vaccination blood samples for testing for which valid results were reported.
Measure: Number; unit: participants
Arm/Group | Arm A: 0.50mL BioThrax, Days 0, 14 | Arm B: 0.50mL BioThrax, Days 0, 28 | Arm C: 0.50mL BioThrax, Days 0, 14, 28 | Arm D: 0.25mL BioThrax, Days 0, 14, 28
Number analyzed (Participants) | 67 | 59 | 59 | 60
participants
  Day 7 | 1 | 0 | 1 | 0
  Day 14 | 4 | 1 | 1 | 0
  Day 21 | 26 | 12 | 19 | 12
  Day 28 | 63 | 13 | 56 | 46
  Day 35 | 65 | 32 | 59 | 53
  Day 42 | 63 | 59 | 59 | 58
  Day 49 | 63 | 59 | 59 | 56
  Day 56 | 59 | 59 | 59 | 55
  Day 63 | 57 | 59 | 59 | 54
  Day 70 | 56 | 59 | 59 | 54
  Day 84 | 44 | 58 | 58 | 51
  Day 100 | 34 | 54 | 56 | 44

2. Secondary Outcome: Geometric Mean Concentration (GMC) of Enzyme-linked Immunosorbent Assay (ELISA) Antibody Against the Protective Antigen (Anti-PA IgG)
Description: Blood was collected from all participants prior to vaccination and at scheduled follow up visits weekly through Day 70, at Day 84 and at Day 100 for testing in the ELISA assay to determine the anti-PA IgG antibody concentration. The geometric mean of subjects' visit-specific titers were calculated along with the 95% confidence intervals. If the antibody titer was below the lower limit of quantification (LLOQ) for the assay, half the value of LLOQ (4.64) was imputed. When all subjects' titers were below LLOQ resulting in no variability within the group, the 95% CI was not calculated.
Time Frame: Days 0, 7, 14, 21, 28, 35, 42, 49, 56, 63, 70, 84 and 100.
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | Arm A: 0.50mL BioThrax, Days 0, 14 | Arm B: 0.50mL BioThrax, Days 0, 28 | Arm C: 0.50mL BioThrax, Days 0, 14, 28 | Arm D: 0.25mL BioThrax, Days 0, 14, 28
Number analyzed (Participants) | 67 | 59 | 59 | 60
µg/mL
  Day 0 | 4.64 [NA to NA] — no variability among the subjects' concentrations | 4.64 [NA to NA] — no variability among the subjects' concentrations | 4.64 [NA to NA] — no variability among the subjects' concentrations | 4.64 [NA to NA] — no variability among the subjects' concentrations
  Day 7 | 5.01 [4.29 to 5.84] | 4.71 [4.56 to 4.86] | 4.91 [4.38 to 5.50] | 4.70 [4.57 to 4.82]
  Day 14 | 6.16 [4.84 to 7.83] | 5.48 [4.85 to 6.18] | 5.28 [4.80 to 5.79] | 5.01 [4.61 to 5.43]
  Day 21 | 13.67 [10.08 to 18.54] | 7.62 [6.18 to 9.41] | 12.11 [9.47 to 15.49] | 7.63 [6.17 to 9.44]
  Day 28 | 88.43 [69.73 to 112.14] | 7.62 [6.22 to 9.33] | 84.05 [67.77 to 104.23] | 52.13 [37.80 to 71.90]
  Day 35 | 89.44 [72.41 to 110.48] | 17.16 [12.34 to 23.87] | 154.49 [125.63 to 189.98] | 86.74 [64.13 to 117.32]
  Day 42 | 76.32 [61.94 to 94.04] | 253.53 [202.43 to 317.52] | 170.40 [140.82 to 206.19] | 108.26 [83.05 to 141.11]
  Day 49 | 61.77 [49.87 to 76.50] | 201.87 [162.54 to 250.73] | 141.93 [117.95 to 170.79] | 93.07 [72.01 to 120.30]
  Day 56 | 52.95 [42.16 to 66.49] | 158.13 [128.27 to 194.95] | 119.28 [98.72 to 144.11] | 77.77 [59.87 to 101.02]
  Day 63 | 41.87 [33.34 to 52.57] | 128.92 [104.68 to 158.76] | 99.20 [82.32 to 119.54] | 66.54 [51.51 to 85.96]
  Day 70 | 36.32 [28.95 to 45.58] | 105.14 [84.81 to 130.35] | 87.13 [72.35 to 104.93] | 56.48 [43.74 to 72.93]
  Day 84 | 25.75 [20.36 to 32.58] | 70.14 [55.63 to 88.44] | 65.42 [54.36 to 78.73] | 43.30 [33.85 to 55.38]
  Day 100 | 19.38 [15.24 to 24.64] | 51.22 [41.48 to 63.23] | 48.77 [40.58 to 58.60] | 32.53 [25.41 to 41.65]

3. Secondary Outcome: Number of Participants Reporting Solicited Injection Site Reactogenicity Symptoms in the Eight Days Following Vaccination at Day 0 by Maximum Severity
Description: Participants maintained a memory aid to record daily the occurrence of local reactions for 8 days after vaccination based on their interference with daily activities (pain, itchiness, warmth, and tenderness at injection site, arm motion limitation) or based on a quantitative measurement of the reaction (edema, erythema). In the subjective grading scale, severe reactions prevented daily activities, moderate reactions interfered with but did not prevent daily activities, and mild reactions did not interfere with daily activities. For the quantitative scale, severe reactions greater than 100 millimeters (mm), moderate reactions were 51-100 mm, and mild reactions were 25-50 mm. Participants are counted by the maximum severity they reported experiencing the reaction on any of the 8 days.
Time Frame: Days 0-7 after vaccination at Day 0
Population: The analysis population includes all participants who were vaccinated at Day 0 per protocol, excluding 59 participants at one clinic site who were vaccinated in the fatty tissue over the triceps rather than the intended inferior deltoid.
Measure: Number; unit: participants
Arm/Group | Arm A: 0.50mL BioThrax, Days 0, 14 | Arm B: 0.50mL BioThrax, Days 0, 28 | Arm C: 0.50mL BioThrax, Days 0, 14, 28 | Arm D: 0.25mL BioThrax, Days 0, 14, 28
Number analyzed (Participants) | 67 | 67 | 68 | 67
participants
  Pain at injection site, severe | 0 | 0 | 0 | 0
  Pain at injection site, moderate | 17 | 12 | 12 | 8
  Pain at injection site, mild | 29 | 41 | 42 | 35
  Itchiness at injection site, severe | 0 | 0 | 0 | 0
  Itchiness at injection site, moderate | 0 | 0 | 1 | 0
  Itchiness at injection site, mild | 11 | 12 | 7 | 10
  Warmth at injection site, severe | 0 | 0 | 0 | 0
  Warmth at injection site, moderate | 2 | 2 | 1 | 2
  Warmth at injection site, mild | 31 | 25 | 28 | 21
  Tenderness at injection site, severe | 0 | 0 | 0 | 0
  Tenderness at injection site, moderate | 22 | 15 | 18 | 10
  Tenderness at injection site, mild | 38 | 44 | 45 | 42
  Arm motion limitations, severe | 0 | 0 | 0 | 0
  Arm motion limitations, moderate | 3 | 4 | 9 | 6
  Arm motion limitations, mild | 14 | 13 | 15 | 10
  Erythema, severe | 0 | 1 | 0 | 0
  Erythema, moderate | 5 | 4 | 5 | 3
  Erythema, mild | 26 | 23 | 21 | 17
  Edema, severe | 0 | 0 | 0 | 0
  Edema, moderate | 4 | 2 | 1 | 1
  Edema, mild | 16 | 17 | 17 | 11

4. Secondary Outcome: Number of Participants Reporting Solicited Injection Site Reactogenicity Symptoms in the Eight Days Following Vaccination at Day 14 by Maximum Severity
Description: as for outcome 3
Time Frame: Days 0-7 after vaccination at Day 14
Population: The analysis population includes all participants who were vaccinated at Day 14 per protocol, excluding 59 participants at one clinic site who were vaccinated in the fatty tissue over the triceps rather than the intended inferior deltoid.
Measure: Number; unit: participants
Arm/Group | Arm A: 0.50mL BioThrax, Days 0, 14 | Arm C: 0.50mL BioThrax, Days 0, 14, 28 | Arm D: 0.25mL BioThrax, Days 0, 14, 28
Number analyzed (Participants) | 65 | 65 | 65
participants
  Pain at injection site, severe | 0 | 0 | 0
  Pain at injection site, moderate | 13 | 12 | 4
  Pain at injection site, mild | 32 | 37 | 35
  Itchiness at injection site, severe | 0 | 0 | 0
  Itchiness at injection site, moderate | 6 | 6 | 3
  Itchiness at injection site, mild | 26 | 21 | 22
  Warmth at injection site, severe | 0 | 0 | 0
  Warmth at injection site, moderate | 4 | 2 | 2
  Warmth at injection site, mild | 30 | 31 | 27
  Tenderness at injection site, severe | 0 | 0 | 0
  Tenderness at injection site, moderate | 24 | 16 | 14
  Tenderness at injection site, mild | 34 | 43 | 43
  Arm motion limitations, severe | 0 | 0 | 0
  Arm motion limitations, moderate | 7 | 2 | 4
  Arm motion limitations, mild | 21 | 20 | 7
  Erythema, severe | 1 | 3 | 0
  Erythema, moderate | 13 | 11 | 9
  Erythema, mild | 19 | 12 | 15
  Edema, severe | 1 | 1 | 0
  Edema, moderate | 10 | 7 | 5
  Edema, mild | 17 | 18 | 11

5. Secondary Outcome: Number of Participants Reporting Solicited Injection Site Reactogenicity Symptoms in the Eight Days Following Vaccination at Day 28 by Maximum Severity
Description: as for outcome 3
Time Frame: Days 0-7 after vaccination at Day 28
Population: The analysis population includes all participants who were vaccinated at Day 28 per protocol, excluding 59 participants at one clinic site who were vaccinated in the fatty tissue over the triceps rather than the intended inferior deltoid.
Measure: Number; unit: participants
Arm/Group | Arm B: 0.50mL BioThrax, Days 0, 28 | Arm C: 0.50mL BioThrax, Days 0, 14, 28 | Arm D: 0.25mL BioThrax, Days 0, 14, 28
Number analyzed (Participants) | 64 | 61 | 61
participants
  Pain at injection site, severe | 0 | 0 | 0
  Pain at injection site, moderate | 11 | 3 | 2
  Pain at injection site, mild | 37 | 24 | 17
  Itchiness at injection site, severe | 0 | 1 | 0
  Itchiness at injection site, moderate | 6 | 3 | 4
  Itchiness at injection site, mild | 21 | 18 | 24
  Warmth at injection site, severe | 0 | 0 | 0
  Warmth at injection site, moderate | 4 | 2 | 1
  Warmth at injection site, mild | 26 | 30 | 27
  Tenderness at injection site, severe | 0 | 1 | 0
  Tenderness at injection site, moderate | 15 | 3 | 4
  Tenderness at injection site, mild | 44 | 43 | 43
  Arm motion limitations, severe | 0 | 0 | 0
  Arm motion limitations, moderate | 3 | 0 | 0
  Arm motion limitations, mild | 16 | 7 | 5
  Erythema, severe | 0 | 1 | 1
  Erythema, moderate | 17 | 6 | 7
  Erythema, mild | 14 | 15 | 17
  Edema, severe | 1 | 0 | 0
  Edema, moderate | 5 | 2 | 5
  Edema, mild | 20 | 13 | 15

6. Secondary Outcome: Number of Participants Reporting Solicited Injection Site Reactogenicity Symptoms in the Eight Days Following the 6-month Boost by Maximum Severity
Description: Participants maintained a memory aid to record daily the occurrence of local reactions for 8 days after the 6-month intramuscular boost vaccination based on their interference with daily activities (pain, itchiness, warmth, and tenderness at injection site, arm motion limitation) or based on a quantitative measurement of the reaction (edema, erythema). In the subjective grading scale, severe reactions prevented daily activities, moderate reactions interfered with but did not prevent daily activities, and mild reactions did not interfere with daily activities. For the quantitative scale, severe reactions greater than 100 millimeters (mm), moderate reactions were 51-100 mm, and mild reactions were 25-50 mm. Participants are counted by the maximum severity they reported experiencing the reaction on any of the 8 days.
Time Frame: Days 0-7 after vaccination at Month 6
Population: The analysis population includes all participants who received the 6-month booster vaccination.
Measure: Number; unit: participants
Arm/Group | Arm A: 0.50mL BioThrax, Days 0, 14 | Arm B: 0.50mL BioThrax, Days 0, 28 | Arm C: 0.50mL BioThrax, Days 0, 14, 28 | Arm D: 0.25mL BioThrax, Days 0, 14, 28
Number analyzed (Participants) | 60 | 60 | 56 | 56
participants
  Pain at injection site, severe | 0 | 1 | 0 | 1
  Pain at injection site, moderate | 20 | 9 | 10 | 13
  Pain at injection site, mild | 24 | 29 | 27 | 20
  Itchiness at injection site, severe | 0 | 0 | 0 | 0
  Itchiness at injection site, moderate | 4 | 2 | 3 | 1
  Itchiness at injection site, mild | 10 | 9 | 6 | 6
  Warmth at injection site, severe | 0 | 0 | 0 | 0
  Warmth at injection site, moderate | 0 | 2 | 4 | 0
  Warmth at injection site, mild | 17 | 17 | 15 | 18
  Tenderness at injection site, severe | 0 | 1 | 0 | 1
  Tenderness at injection site, moderate | 16 | 9 | 15 | 14
  Tenderness at injection site, mild | 33 | 42 | 28 | 30
  Arm motion limitations, severe | 0 | 0 | 0 | 1
  Arm motion limitations, moderate | 7 | 6 | 7 | 9
  Arm motion limitations, mild | 16 | 8 | 14 | 13
  Erythema, severe | 0 | 0 | 1 | 0
  Erythema, moderate | 1 | 3 | 0 | 1
  Erythema, mild | 4 | 1 | 5 | 1
  Edema, severe | 0 | 0 | 0 | 0
  Edema, moderate | 3 | 2 | 1 | 2
  Edema, mild | 5 | 2 | 2 | 2

7. Secondary Outcome: Number of Participants With Injection Site Edema and Erythema With a Size of Greater Than 120 Millimeters (mm)
Description: Participants were given a ruler with the memory aid to measure the occurrence of edema (swelling) and erythema (redness) daily for at least 8 days after each vaccination. Participants are counted in this outcome measure if they had measurements of greater than 120 mm in the 8-day period after at least one vaccination, first separately for edema and erythema, and in the last category, edema and/or erythema, if they had either or both reactions of greater than 120 mm.
Time Frame: Days 0-7 after each vaccination
Population: The analysis population includes all participants who were vaccinated per protocol, excluding 59 participants at one clinic site who were vaccinated in the fatty tissue over the triceps rather than the intended inferior deltoid.
Measure: Number; unit: participants
Arm/Group | Arm A: 0.50mL BioThrax, Days 0, 14 | Arm B: 0.50mL BioThrax, Days 0, 28 | Arm C: 0.50mL BioThrax, Days 0, 14, 28 | Arm D: 0.25mL BioThrax, Days 0, 14, 28
Number analyzed (Participants) | 67 | 67 | 68 | 67
participants
  Edema | 1 | 1 | 1 | 0
  Erythema | 1 | 1 | 2 | 1
  Edema and/or Erythema | 1 | 2 | 2 | 1

8. Secondary Outcome: TNA NF50 Geometric Mean Titers (GMT) at Days 0, 7, 14, 21, 28, 35, 42, 49, 56, 63, 70, 84 and 100.
Description: Blood was collected from all participants prior to vaccination and at scheduled follow up visits weekly through Day 70, at Day 84 and at Day 100 for testing in the toxin neutralization antibody assay to determine the NF50 antibody titer. The geometric mean of subjects' visit-specific titers were calculated along with the 95% confidence intervals. If the antibody titer was below the lower limit of quantification (LLOQ) for the assay, half the value of LLOQ (0.03) was imputed. When all subjects' titers were below LLOQ resulting in no variability within the group, the 95% CI was not calculated.
Time Frame: Days 0, 7, 14, 21, 28, 35, 42, 49, 56, 63, 70, 84 and 100.
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Arm A: 0.50mL BioThrax, Days 0, 14 | Arm B: 0.50mL BioThrax, Days 0, 28 | Arm C: 0.50mL BioThrax, Days 0, 14, 28 | Arm D: 0.25mL BioThrax, Days 0, 14, 28
Number analyzed (Participants) | 67 | 59 | 59 | 60
titer
  Day 0 | 0.03 [NA to NA] — no variability among the subjects' titers | 0.03 [NA to NA] — no variability among the subjects' titers | 0.03 [NA to NA] — no variability among the subjects' titers | 0.03 [NA to NA] — no variability among the subjects' titers
  Day 7 | 0.03 [0.03 to 0.04] | 0.03 [NA to NA] — no variability among the subjects' titers | 0.03 [0.03 to 0.04] | 0.03 [NA to NA] — no variability among the subjects' titers
  Day 14 | 0.04 [0.03 to 0.05] | 0.04 [0.03 to 0.04] | 0.04 [0.03 to 0.04] | 0.03 [0.03 to 0.03]
  Day 21 | 0.10 [0.07 to 0.13] | 0.06 [0.04 to 0.08] | 0.08 [0.06 to 0.11] | 0.05 [0.04 to 0.07]
  Day 28 | 0.62 [0.48 to 0.80] | 0.06 [0.05 to 0.08] | 0.65 [0.50 to 0.85] | 0.38 [0.26 to 0.55]
  Day 35 | 0.61 [0.49 to 0.76] | 0.17 [0.12 to 0.24] | 1.22 [0.98 to 1.51] | 0.75 [0.55 to 1.02]
  Day 42 | 0.51 [0.41 to 0.63] | 2.85 [2.21 to 3.67] | 1.33 [1.09 to 1.62] | 0.91 [0.70 to 1.18]
  Day 49 | 0.41 [0.33 to 0.50] | 2.19 [1.74 to 2.76] | 1.02 [0.84 to 1.24] | 0.74 [0.57 to 0.98]
  Day 56 | 0.35 [0.28 to 0.44] | 1.62 [1.28 to 2.04] | 0.83 [0.68 to 1.02] | 0.61 [0.47 to 0.80]
  Day 63 | 0.27 [0.21 to 0.33] | 1.27 [1.00 to 1.62] | 0.71 [0.58 to 0.86] | 0.51 [0.39 to 0.67]
  Day 70 | 0.24 [0.19 to 0.29] | 1.00 [0.79 to 1.26] | 0.60 [0.49 to 0.73] | 0.44 [0.34 to 0.57]
  Day 84 | 0.17 [0.13 to 0.21] | 0.64 [0.51 to 0.81] | 0.45 [0.37 to 0.54] | 0.30 [0.23 to 0.39]
  Day 100 | 0.13 [0.10 to 0.16] | 0.44 [0.35 to 0.55] | 0.34 [0.28 to 0.41] | 0.24 [0.18 to 0.30]

9. Secondary Outcome: Peak Geometric Mean Concentration (GMC) of ELISA Anti-PA IgG Antibody Through Day 100
Description: Blood was collected from all participants prior to vaccination and at scheduled follow up visits weekly through Day 70, at Day 84 and at Day 100 for testing in the ELISA assay to determine the anti-PA IgG antibody concentration. To determine the group peak GMC, the highest antibody concentration assessed for each subject at any post vaccination visit through Day 100 was determined. The geometric mean of subjects' peak concentrations was calculated along with the 95% confidence intervals.
Time Frame: Day 7 through Day 100
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | Arm A: 0.50mL BioThrax, Days 0, 14 | Arm B: 0.50mL BioThrax, Days 0, 28 | Arm C: 0.50mL BioThrax, Days 0, 14, 28 | Arm D: 0.25mL BioThrax, Days 0, 14, 28
Number analyzed (Participants) | 67 | 59 | 59 | 60
µg/mL | 102.32 [82.31 to 127.19] | 265.08 [214.11 to 328.18] | 182.42 [150.28 to 221.42] | 114.42 [87.49 to 149.64]

10. Secondary Outcome: Number of Participants Reporting Solicited Subjective Systemic Symptoms for Eight Days After Vaccination at Day 0 by Maximum Severity.
Description: Participants maintained a memory aid to record daily the occurrence of solicited systemic reactions of fatigue, muscle aches, and headache for 8 days after vaccination based on their interference with daily activities. Severe reactions prevented daily activities, moderate reactions interfered with but did not prevent daily activities, and mild reactions did not interfere with daily activities. Participants are counted by the maximum severity they reported experiencing the reaction on any of the 8 days.
Time Frame: Days 0-7 after vaccination at Day 0
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Arm A: 0.50mL BioThrax, Days 0, 14 | Arm B: 0.50mL BioThrax, Days 0, 28 | Arm C: 0.50mL BioThrax, Days 0, 14, 28 | Arm D: 0.25mL BioThrax, Days 0, 14, 28
Number analyzed (Participants) | 67 | 67 | 68 | 67
participants
  Fatigue, severe | 0 | 0 | 0 | 0
  Fatigue, moderate | 6 | 6 | 8 | 3
  Fatigue, mild | 9 | 12 | 12 | 15
  Muscle aches, severe | 0 | 0 | 0 | 0
  Muscle aches, moderate | 2 | 2 | 7 | 4
  Muscle aches, mild | 15 | 16 | 12 | 14
  Headache, severe | 0 | 0 | 0 | 0
  Headache, moderate | 6 | 3 | 4 | 3
  Headache, mild | 9 | 13 | 15 | 18

11. Secondary Outcome: Number of Participants Reporting Solicited Subjective Systemic Symptoms for Eight Days After Vaccination at Day 14 by Maximum Severity.
Description: as for outcome 10
Time Frame: Days 0-7 after vaccination at Day 14
Population: as for outcome 4
Measure: Number; unit: participants
Arm/Group | Arm A: 0.50mL BioThrax, Days 0, 14 | Arm C: 0.50mL BioThrax, Days 0, 14, 28 | Arm D: 0.25mL BioThrax, Days 0, 14, 28
Number analyzed (Participants) | 65 | 65 | 65
participants
  Fatigue, severe | 0 | 0 | 0
  Fatigue, moderate | 7 | 3 | 5
  Fatigue, mild | 17 | 15 | 10
  Muscle aches, severe | 0 | 0 | 0
  Muscle aches, moderate | 7 | 6 | 3
  Muscle aches, mild | 18 | 13 | 14
  Headache, severe | 0 | 0 | 0
  Headache, moderate | 4 | 4 | 4
  Headache, mild | 14 | 17 | 11

12. Secondary Outcome: Number of Participants Reporting Solicited Subjective Systemic Symptoms for Eight Days After Vaccination at Day 28 by Maximum Severity.
Description: as for outcome 10
Time Frame: Days 0-7 after vaccination at Day 28
Population: as for outcome 5
Measure: Number; unit: participants
Arm/Group | Arm B: 0.50mL BioThrax, Days 0, 28 | Arm C: 0.50mL BioThrax, Days 0, 14, 28 | Arm D: 0.25mL BioThrax, Days 0, 14, 28
Number analyzed (Participants) | 64 | 61 | 61
participants
  Fatigue, severe | 0 | 0 | 1
  Fatigue, moderate | 2 | 2 | 0
  Fatigue, mild | 10 | 7 | 13
  Muscle aches, severe | 0 | 0 | 0
  Muscle aches, moderate | 3 | 3 | 0
  Muscle aches, mild | 14 | 7 | 12
  Headache, severe | 0 | 0 | 0
  Headache, moderate | 3 | 0 | 1
  Headache, mild | 8 | 8 | 12

13. Secondary Outcome: Number of Participants Reporting Solicited Subjective Systemic Symptoms for Eight Days After the 6-month Boost Vaccination by Maximum Severity.
Description: Participants maintained a memory aid to record daily the occurrence of solicited systemic reactions of fatigue, muscle aches, and headache for 8 days after the 6-month intramuscular boost vaccination based on their interference with daily activities. Severe reactions prevented daily activities, moderate reactions interfered with but did not prevent daily activities, and mild reactions did not interfere with daily activities. Participants are counted by the maximum severity they reported experiencing the reaction on any of the 8 days.
Time Frame: Days 0-7 after vaccination at Month 6
Population: The analysis population includes all participants who received the 6-month boost vaccination.
Measure: Number; unit: participants
Arm/Group | Arm A: 0.50mL BioThrax, Days 0, 14 | Arm B: 0.50mL BioThrax, Days 0, 28 | Arm C: 0.50mL BioThrax, Days 0, 14, 28 | Arm D: 0.25mL BioThrax, Days 0, 14, 28
Number analyzed (Participants) | 60 | 60 | 56 | 56
participants
  Fatigue, severe | 0 | 0 | 0 | 0
  Fatigue, moderate | 6 | 2 | 3 | 1
  Fatigue, mild | 9 | 10 | 13 | 13
  Muscle aches, severe | 0 | 0 | 0 | 0
  Muscle aches, moderate | 8 | 2 | 6 | 4
  Muscle aches, mild | 13 | 14 | 14 | 15
  Headache, severe | 0 | 0 | 0 | 0
  Headache, moderate | 7 | 0 | 4 | 1
  Headache, mild | 3 | 7 | 9 | 6

14. Secondary Outcome: Number of Participants Reporting Fever in the Eight Days After Vaccination at Day 0 by Maximum Severity
Description: Participants were given a thermometer with a memory aid to record their oral temperature at least once daily, encouraged to be at the same time each day, but at any time the participant felt they may have a fever. The highest temperature assessed for each day was reported and graded according to the protocol grading scale of severe being greater than or equal to 39 degrees Celsius, moderate 38.5-38.9 degrees Celsius, and mild 38.0-38.4 degrees Celsius. Participants are counted by the maximum severity they reported experiencing fever on any of the 8 days.
Time Frame: Day 0-7 after vaccination at Day 0
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Arm A: 0.50mL BioThrax, Days 0, 14 | Arm B: 0.50mL BioThrax, Days 0, 28 | Arm C: 0.50mL BioThrax, Days 0, 14, 28 | Arm D: 0.25mL BioThrax, Days 0, 14, 28
Number analyzed (Participants) | 67 | 66 | 68 | 67
participants
  Fever, severe | 0 | 0 | 0 | 0
  Fever, moderate | 0 | 0 | 0 | 0
  Fever, mild | 0 | 0 | 0 | 0

15. Secondary Outcome: Number of Participants Reporting Fever in the Eight Days After Vaccination at Day 14 by Maximum Severity
Description: as for outcome 14
Time Frame: Day 0-7 after vaccination at Day 14
Population: as for outcome 4
Measure: Number; unit: participants
Arm/Group | Arm A: 0.50mL BioThrax, Days 0, 14 | Arm C: 0.50mL BioThrax, Days 0, 14, 28 | Arm D: 0.25mL BioThrax, Days 0, 14, 28
Number analyzed (Participants) | 65 | 65 | 65
participants
  Fever, severe | 0 | 0 | 0
  Fever, moderate | 0 | 0 | 0
  Fever, mild | 0 | 0 | 0

16. Secondary Outcome: Number of Participants Reporting Fever in the Eight Days After Vaccination at Day 28 by Maximum Severity
Description: as for outcome 14
Time Frame: Day 0-7 after vaccination at Day 28
Population: as for outcome 5
Measure: Number; unit: participants
Arm/Group | Arm B: 0.50mL BioThrax, Days 0, 28 | Arm C: 0.50mL BioThrax, Days 0, 14, 28 | Arm D: 0.25mL BioThrax, Days 0, 14, 28
Number analyzed (Participants) | 64 | 60 | 61
participants
  Fever, severe | 0 | 0 | 0
  Fever, moderate | 0 | 0 | 0
  Fever, mild | 0 | 0 | 0

17. Secondary Outcome: Number of Participants Reporting Fever in the Eight Days After the 6-month Boost Vaccination by Maximum Severity
Description: as for outcome 14
Time Frame: Day 0-7 after vaccination at Month 6
Population: The analysis population includes all participants who received the 6-month boost vaccination and recorded oral temperatures.
Measure: Number; unit: participants
Arm/Group | Arm A: 0.50mL BioThrax, Days 0, 14 | Arm B: 0.50mL BioThrax, Days 0, 28 | Arm C: 0.50mL BioThrax, Days 0, 14, 28 | Arm D: 0.25mL BioThrax, Days 0, 14, 28
Number analyzed (Participants) | 60 | 58 | 55 | 56
participants
  Fever, severe | 0 | 0 | 1 | 0
  Fever, moderate | 0 | 0 | 0 | 0
  Fever, mild | 0 | 0 | 0 | 1

18. Secondary Outcome: Number of Subjects With a Four-fold or Greater Increase From Baseline in Enzyme-linked Immunosorbent Assay (ELISA) Antibody Concentration Against the Protective Antigen (Anti-PA IgG)
Description: Blood was collected from all participants prior to vaccination and at scheduled follow up visits weekly through Day 70, at Day 84 and at Day 100 for testing in the ELISA assay to determine the anti-PA IgG antibody concentration. A participant met the threshold of a 4-fold rise in anti-PA IgG antibody concentration if the post vaccination concentration was an increase by 4-fold or more from the baseline (Day 0) concentration.
Time Frame: Days 0, 7, 14, 21, 28, 35, 42, 49, 56, 63, 70, 84 and 100.
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Arm A: 0.50mL BioThrax, Days 0, 14 | Arm B: 0.50mL BioThrax, Days 0, 28 | Arm C: 0.50mL BioThrax, Days 0, 14, 28 | Arm D: 0.25mL BioThrax, Days 0, 14, 28
Number analyzed (Participants) | 67 | 59 | 59 | 60
participants
  Day 7 | 1 | 0 | 1 | 0
  Day 14 | 4 | 2 | 0 | 1
  Day 21 | 25 | 9 | 21 | 11
  Day 28 | 65 | 9 | 57 | 46
  Day 35 | 65 | 24 | 59 | 54
  Day 42 | 65 | 59 | 59 | 57
  Day 49 | 61 | 59 | 59 | 56
  Day 56 | 60 | 59 | 59 | 55
  Day 63 | 57 | 59 | 59 | 53
  Day 70 | 54 | 58 | 58 | 53
  Day 84 | 44 | 56 | 57 | 49
  Day 100 | 38 | 52 | 54 | 48

19. Secondary Outcome: TNA NF50 Peak Geometric Mean Titer (GMT) Antibody Response Through Day 100
Description: Blood was collected from all participants prior to vaccination and at scheduled follow up visits weekly through Day 70, at Day 84 and at Day 100 for testing in the toxin neutralization antibody assay to determine the NF50 antibody titer. To determine the group peak GMT, the highest titer assessed for each subject at any post vaccination visit through Day 100 was determined. The geometric mean of each subjects' peak titers was calculated along with the 95% confidence intervals.
Time Frame: Day 7 through Day 100
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Arm A: 0.50mL BioThrax, Days 0, 14 | Arm B: 0.50mL BioThrax, Days 0, 28 | Arm C: 0.50mL BioThrax, Days 0, 14, 28 | Arm D: 0.25mL BioThrax, Days 0, 14, 28
Number analyzed (Participants) | 67 | 59 | 59 | 60
titer | 0.74 [0.59 to 0.94] | 2.99 [2.34 to 3.81] | 1.48 [1.22 to 1.81] | 1.00 [0.76 to 1.32]

ADVERSE EVENTS:
Time Frame: Solicited events were collected for 8 days after each vaccination, unsolicited AEs through 28 days after last vaccination in the primary series and 21 days after the boost vaccination, and serious adverse events through 201 days after first vaccination.
Description: For events solicited on a Memory Aid in the 8 days after vaccination, a participant was considered to have one event if it was reported as experienced at any time in the 8-day period. Each 8-day period was considered a separate event.
Arm/Group | Arm A: 0.50mL BioThrax, Days 0, 14 | Arm B: 0.50mL BioThrax, Days 0, 28 | Arm C: 0.50mL BioThrax, Days 0, 14, 28 | Arm D: 0.25mL BioThrax, Days 0, 14, 28
Serious Adverse Events (participants affected / at risk) | 0/82 | 2/82 | 1/82 | 0/82
Other Adverse Events (participants affected / at risk) | 82/82 | 82/82 | 82/82 | 82/82
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: 0.50mL BioThrax, Days 0, 14 (N=82) | Arm B: 0.50mL BioThrax, Days 0, 28 (N=82) | Arm C: 0.50mL BioThrax, Days 0, 14, 28 (N=82) | Arm D: 0.25mL BioThrax, Days 0, 14, 28 (N=82)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Localised infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Convulsion (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: 0.50mL BioThrax, Days 0, 14 (N=82) | Arm B: 0.50mL BioThrax, Days 0, 28 (N=82) | Arm C: 0.50mL BioThrax, Days 0, 14, 28 (N=82) | Arm D: 0.25mL BioThrax, Days 0, 14, 28 (N=82)
Fatigue (General disorders) | 38 (58) | 33 (48) | 40 (74) | 40 (70)
Myalgia (Musculoskeletal and connective tissue disorders) | 47 (75) | 35 (58) | 38 (75) | 42 (75) — Solicited as 'muscle aches' on the memory aid
Headache (Nervous system disorders) | 32 (49) | 30 (44) | 42 (68) | 40 (66)
Vaccination site pain (General disorders) | 71 (155) | 72 (168) | 72 (185) | 71 (154)
Vaccination site pruritus (General disorders) | 52 (74) | 44 (64) | 47 (81) | 48 (88)
Vaccination site warmth (General disorders) | 54 (102) | 49 (88) | 50 (124) | 50 (120)
Tenderness (General disorders) | 81 (205) | 79 (208) | 80 (251) | 78 (247)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 44 (79) | 39 (59) | 48 (85) | 43 (63) — Solicited as "arm motion limitations" on the memory aid
Vaccination site erythema (General disorders) | 53 (84) | 48 (86) | 47 (91) | 42 (94)
Vaccination site swelling (General disorders) | 44 (74) | 44 (63) | 40 (73) | 40 (70)
Bradycardia (Cardiac disorders) | 2 (2) | 4 (4) | 8 (11) | 7 (11)
Dizziness (Nervous system disorders) | 0 (0) | 2 (2) | 4 (5) | 5 (5)
Headache (Nervous system disorders) | 7 (8) | 5 (6) | 5 (6) | 4 (4)
Hypertension (Vascular disorders) | 1 (1) | 4 (7) | 5 (7) | 2 (4)
Nasopharyngitis (Infections and infestations) | 5 (5) | 6 (6) | 5 (5) | 6 (6)
Respiratory rate increased (Investigations) | 21 (27) | 25 (34) | 26 (37) | 22 (30)
Upper respiratory tract infection (Infections and infestations) | 9 (9) | 18 (19) | 13 (14) | 10 (11)
Vaccination site bruising (General disorders) | 6 (6) | 10 (12) | 4 (4) | 5 (5)
Vaccination site erythema (General disorders) | 4 (4) | 6 (7) | 4 (4) | 3 (3) — Vaccination site erythema that persisted beyond 14 days post vaccination was reported as an unsolicited adverse event.
Vaccination site nodule (General disorders) | 63 (109) | 64 (107) | 66 (145) | 60 (129)
Vessel puncture site bruise (General disorders) | 5 (5) | 2 (2) | 3 (3) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less